CLINICAL TRIAL: NCT06958770
Title: Combining Electrical Impedance Tomography and Thoracic Ultrasound to Investigate Dynamic Changes of Respiratory Effort, and Regional & End-expiratory Lung Volume in Mechanically Ventilated Patients.
Brief Title: Combining Electrical Impedance Tomography and Thoracic Ultrasound Toinvestigate Dynamic Changes
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202502091RIND
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: ARDS (Moderate or Severe)
Keywords: Chest ultrasound; electrical impedance tomography
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Oxygen Consumption

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electrical impedance tomography — * Electrical impedance tomography (EIT)：Assessing pulmonary function in chronic lung diseases.
  * Lung ultrasound：Assessing diaphragm atrophy in mechanically ventilated patients.
  * Esophageal pressure：The work of breathing, or the energy required by respiratory muscles to meet ventilatory demands, can be directly evaluated by esophageal pressure
  * Oxygen consumption：Indirectly evaluated by measuring oxygen consumption (V̇O2) during mechanical ventilation The oxygen cost of breathing, reflected the increase in V̇O2 when transitioning from mechanical ventilation to spontaneous breathing, has been shown to predict weaning outcomes.
  Other Names: Lung ultrasound; Esophageal pressure; Oxygen consumption

SUMMARY:
1. To evaluate the dynamic changes of lung ultrasound during electrical impedance tomography (EIT) PEEP titration and across the first week of ARDS.
2. To asses respiratory effort by diaphragmatic function, esophageal pressure, and EIT (Pendelluft phenomenon), and hyperinflammatory biomarkers, to predict P-SILI.
3. To develop predictive models for weaning success based on integrated EELI and thoracic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 y/o.
* Patient intubated and receiving mechanical ventilation > 24 hours.
* Admitted into ICU, diagnosed as moderate or severe ARDS (ICD-10-CM: J80) according to Berlin definition.

Exclusion Criteria:

* Presence of Implanted Electronic Devices (pacemakers, implantable cardioverter-defibrillators).
* Pregnancy.
* No consent/inability to obtain consent and appropriate legal representative not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted into ICU, diagnosed as moderate or severe ARDS (ICD-10-CM: J80) according to Berlin definition.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ARDS | From enrollment to the end of treatment at 1 weeks.
  Correlation of LUS aeration scores and overdistension metrics (e.g., A-line prominence, reduced lung sliding) with EIT parameters, including hyperdistension (%), collapse (%), and ΔEELI.
  Correlation of P-SILI risk with diaphragmatic function (ultrasound-measured excursion and thickening fraction), esophageal pressure variations (ΔPes, ΔPdi), pendelluft dynamics (phase shift, amplitude difference from EIT), and hyperinflammatory biomarkers (e.g., IL-6, IL-8).

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No